CLINICAL TRIAL: NCT07214129
Title: Safety and Efficacy of Nebulized Nitroglycerin as a Vaso-reactive Agent in Pulmonary Arterial Hypertension
Brief Title: Safety and Efficacy of Nebulized Nitroglycerin in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD.22.02.608.R1
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Nebulized nitroglycerin; pulmonary arterial hypertension; vaso-reactive agent
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pulmonary arterial hypertension patients received Nebulized nitroglycerin as a vaso-reactive agent (Experimental): A local anesthetic is administered subcutaneously at the access site. Venous access is obtained with or without ultrasound guidance. Once venous access is obtained, an appropriately sized sheath is placed in the vein and secured. The pulmonary artery catheter is advanced through the sheath into the vein. The balloon is inflated after the catheter is advanced to roughly 15 cm so to avoid inflating it within the access sheath. Balloon inflation will then make advancing the catheter to the right atrium much easier.
  The catheter movement will be monitored by changes in wave forms or observed using fluoroscopy.
  Prior to recording pressures, a reference will be established by zeroing the system. Zeroing involves opening the air-fluid transducer to air so that it equilibrates with atmospheric pressure.
  After obtaining hemodynamic data, nitroglycerin inhalation will be given at dose 5 mg via nebulizer device over 15 minutes then reassessment will be carried out.
  Interventions: Drug: Nebulized nitroglycerin

INTERVENTIONS:
Drug: Nebulized nitroglycerin — Nebulized nitroglycerin as vaso-reactive agen in pulmonary arterial hypertension
  Other Names: Nitroglycerin

SUMMARY:
The 6th World Symposium on Pulmonary Hypertension, pre-capillary pulmonary hypertension (PH) has been defined as mean pulmonary arterial pressure (mPAP) >20 mm Hg with a pulmonary arterial wedge pressure (PAWP) ≤15 mm Hg and pulmonary vascular resistance (PVR) ≥3 Wood units (WU). The current classification of PH categorizes clinical conditions associated with PH based on similar pathophysiology, etiologies, clinical presentation, hemodynamic characteristics and therapeutic management. PH is classified into five groups. The group 1 pulmonary arterial hypertension (PAH), which comprises of diverse diseases that result in similar pathological changes within the pulmonary vasculature. This includes idiopathic, familial, drug and toxin induced PAH and associated forms of PAH like systemic sclerosis, portal hypertension, congenital heart disease and human immunodeficiency virus (HIV). The remaining 4 groups of PH are secondary to other conditions and are usually referred to as secondary PH

DETAILED DESCRIPTION:
Right Heart Catheterization (RHC) is the diagnostic gold standard for pulmonary hypertension (PH), In fact, RHC is the definitive diagnostic technique for reliably confirming whether a patient has PAH .In addition to its use in diagnosis, RHC provides useful information on the degree of hemodynamic impairment, determines response to PAH therapy and establishes prognosis, thereby informing clinical decision-making in the management of PAH. Acute vaso-reactivity test (AVT) is defined as "a fall of at least 10 mmHg in mean pulmonary artery pressure (PAP); a fall to an absolute mean PAP less than 40 mmHg; and unchanged or increased cardiac output". AVT is typically performed with a short-acting agent such as inhaled nitric oxide, inhaled iloprost, intravenous epoprostenol, or adenosine. Baseline hemodynamic measurements are obtained prior to testing. AVT is performed for three reasons in pulmonary hypertension (PH): 1) identification of patients who may display a favorable long-term response to calcium channel blocker treatment, 2) gathering prognostic information,3) scientific research purposes.

The aim of this study is to evaluate the safety and efficacy of nebulized nitroglycerin as a vaso-reactive agent in pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with clinical and echocardiographic features suggestive of pulmonary hypertension after exclusion of all secondary causes.

Exclusion Criteria:

* groups 2,3,4,5 Pulmonary hypertension
* Hemodynamic instability.
* Absolute contraindications to pulmonary artery catheter (PAC) placement include: Infection at the insertion site The presence of a right ventricular assist device Insertion during cardiopulmonary bypass Lack of consent
* Relative contraindications to the placement of a PAC include a coagulopathy (international normalized ratio >1.5), thrombocytopenia (platelet count <50,000/microL), electrolyte disturbances (hypo- or hyper-kalemia, -magnesemia, -natremia, -calcemia), and severe acid-base disturbances (eg, pH <7.2 or >7.5).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Nebulized nitroglycerin as vaso-reactive agent in pulmonary arterial hypertension | 6 months
  Nebulized nitroglycerin cause vasodilation in pulmonary arterial hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt